CLINICAL TRIAL: NCT03729102
Title: Immunological Tolerance After Frequent Rabies Booster Vaccinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal Investigator, Queen Saovabha Memorial Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QSMI-IRB 2/2018
Record Dates: First submitted 2018-10-30; First posted 2018-11-02 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Rabies
Keywords: rabies vaccination
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Intervention Model Description: There would be two study groups. Those who had received primary immunization would be the control group. While persons who had received primary immunization and later received booster vaccination for at least 3 times would be the study group.
  All participants would be given one dose of rabies vaccine and monitored the immunological cells and cytokines before and after the rabies booster injection.
Who Masked: Outcomes Assessor
Masking Description: The serum samples from all participants would be labelled as the codes, of which the laboratory technicians could not access to the groups or other details of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Persons who had received primary immunization
  Interventions: Biological: Blood drawn after rabies vaccine booster vaccination
- Study group (Experimental): Persons who had received primary immunization and later received booster vaccination for at least 3 times
  Interventions: Biological: Blood drawn after rabies vaccine booster vaccination

INTERVENTIONS:
Biological: Blood drawn after rabies vaccine booster vaccination — All participants would be given one dose of rabies vaccine and monitor the immunological cells i.e., regulatory T cell, regulatory B cell, T follicular helper cells, cytokines i.e., IL-10, TGF-Beta, and Rabies neutralizing antibody titers, before and after the booster injection

SUMMARY:
To study immunological tolerance effect after frequent rabies booster vaccination

DETAILED DESCRIPTION:
Previous studies had shown lower antibody titers among those who received frequent rabies booster vaccination, compared to ones who had got primary immunization. We study immunological cells i.e., regulatory T cell, regulatory B cell, T follicular helper cell, and cytokines in those who received frequent rabies booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Previously received rabies vaccination

Exclusion Criteria:

* Had immunocompromised conditions
* Received blood or blood product within 3 months
* Received anti-malarial drugs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rabies specific regulatory T cells | Change from baseline of numbers of Rabies specific regulatory T cells before (baseline) and one month after receipt of rabies booster vaccination were compared between 2 arms
  Rabies specific regulatory T cells are measured by flow cytometry method
Rabies specific regulatory B cells | Change from baseline of numbers of Rabies specific regulatory B cells before (baseline) and one month after receipt of rabies booster vaccination were compared between 2 arms
  Rabies specific regulatory B cells are measured by flow cytometry method
Rabies specific T follicular helper cells | Change from baseline of numbers of Rabies specific T follicular helper cells before (baseline) and one month after receipt of rabies booster vaccination were compared between 2 arms
  Rabies specific T follicular helper cells are measured by flow cytometry method

SECONDARY OUTCOMES:
Rabies Neutralizing Antibody Titers (RNab) | before (baseline) and one month after receipt of rabies booster vaccination
  Rabies Neutralizing Antibody Titers would be represented and compared by geometric mean titers (GMTs)

OTHER OUTCOMES:
Cytokines | Change from baseline of quantitative measurement of cytokines levels would be measured before (baseline) and one month after receipt of rabies booster vaccination and compared between 2 arms
  Cytokines i.e., IL-10, TGF-Beta are measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No